CLINICAL TRIAL: NCT05830422
Title: Prediction of Delayed Cognitive Impairment in Cardiac Arrest Survivors With Good Neurological Outcomes
Status: Enrolling by invitation | Type: Observational
Sponsor: Chungnam National University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CNUH 2022-10-059-004
Record Dates: First submitted 2023-03-29; First posted 2023-04-26 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2023-03

CONDITIONS: Cardiac Arrest, Out-Of-Hospital; Cognitive Impairment
Keywords: cardiac arrest; outcome; cognition impairment; magnetic resonance imaging; Positron emission tomography
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Cognitive Dysfunction; Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — Blood was collected 10-14 days, 3 months, and 6 months after ROSC by venipuncture, and the obtained blood was collected in an SST bottle without anticoagulant and centrifuged (3,000 rpm, 10 minutes or more) within 60 minutes. Divided into tubes, and pre-treated tubes are stored frozen at -70 degrees.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Good neurological outcome: Patients who showed good neurological outcomes with CPC scores of 1-2 at discharge
  Interventions: Other: nothing

INTERVENTIONS:
Other: nothing — Follow-up observation was conducted without any intervention in an outpatient setting.

SUMMARY:
The objective of this observational study is to provide basic data for predicting and analyzing the occurrence and causes of delayed cognitive impairment, an important factor in the quality of life, among discharged patients who have received targeted temperature management therapy and experienced favorable neurological outcomes after out-of-hospital cardiac arrest.

The main questions it aims to answer are:

* Can we identify abnormal areas in the brains of patients with delayed cognitive impairment using Brain MRI or positron emission tomography (PET) imaging?
* Is it possible to predict delayed cognitive impairment using biomarkers?

DETAILED DESCRIPTION:
1. For study subjects who survived after out-of-hospital cardiac arrest, prognosis was evaluated using Cerebral Performance Category (CPC) scores on days 10-14 after return of spontaneous circulation (ROSC). A CPC score of 1-2 indicates a good neurological prognosis, while a score of 3-5 indicates a poor neurological prognosis. Only subjects with CPC scores of 1-2 were included in this study.
2. Blood samples were collected through venous puncture at days 10-14, 3 months, and 6 months after ROSC, and the obtained blood was drawn into an serum separating tube (SST) bottle without anticoagulants, then centrifuged within 60 minutes after collection (at 3,000rpm for at least 10 minutes) and divided into tubes. The processed tubes were stored at -70°C.

   * The storage period of the samples is 5 years from the date of collection, and they are stored in a coded manner for anonymization.
   * The Human Neurology 4-ples A 2.0 Assay Kit (including neurofilament light chain, Tau protein, ubiquitin carboxyl terminal esterase L1 protein [UCHL1], and glial fibrillary acidic protein antibody) was analyzed using the single molecule protein detection (SIMOA) analysis machine, and neuron-specific enolase (NSE) in the blood was analyzed together as a reference point to assess the usefulness of each biomarker.
3. Through the Seoul Neuropsychological Screening Battery (SNSB), attention, language and related functions, visuospatial function, memory, frontal lobe and executive function, and other related functions can be assessed. The test is conducted by a specialist clinical psychologist for 1 hour and 30 minutes to 2 hours, and the results are analyzed by Professor Oh Eung-Seok, a neurologist. The presence of cognitive impairment is assessed by conducting tests at 10-14 days, 3 months, and 6 months after ROSC for out-of-hospital cardiac arrest patients with CPC 1-2 points who have passed 10-14 days since ROSC. In addition, through detailed item analysis of the SNSB, functional abnormalities and affected areas (such as the frontal lobe, parietal lobe, temporal lobe, and occipital lobe) are analyzed.
4. We consulted with the departments of radiology, nuclear medicine, and neurology professors to establish the optimal fluorine-18 (18F) fluorodeoxyglucose (FDG) PET & MRI examination protocol. The first MRI examination was performed 72-96 hours after ROSC, as recommended by international treatment guidelines for predicting neurological prognosis. The first [18F]-FDG PET examination was performed at 10-14 days after ROSC, as it may result in false positives if performed too early in cardiac arrest patients. A minimum of 10 days is recommended before performing the examination. If cognitive impairment is observed in the SNSB examination at 3 months after ROSC, a second [18F]-FDG PET & MRI examination is performed. If the cognitive function is normal at 6 months, the examination is performed regardless of cognitive impairment.
5. Prediction and analysis of delayed cognitive impairment and cause analysis in out-of-hospital cardiac arrest patients with good neurological outcomes
6. Delayed cognitive impairment is defined based on the SNSB results, and is defined as the positive group. For biomarkers, differences between the positive and negative groups are determined at each time point, and the predictive power and cut-off values are determined using area under the receiver operating characteristics curve. For images, the functional or anatomical differences between the two groups are compared.
7. Predictive power analysis Through SNSB, the patient's cognitive impairment and the time point of recognition are measured, and the level of biomarkers tested prior to the recognition of impairment is checked to analyze the predictive power. Therefore, the time points for predictive power analysis are 10-14 days, 3 months, and 6 months after ROSC. The first and second [18F]-FDG PET & MRI findings are analyzed to identify differences between the cognitive impairment group and the normal group. Using multiple modes combining clinical data, biomarkers, [18F]-FDG PET, MRI, etc., a predictive model for delayed cognitive impairment is developed.
8. Cause analysis Investigate the impairment findings and location using the continuously measured SNSB test values. Analyze the first and second [18F]-FDG PET and MRI findings to investigate the functional or anatomical abnormalities occurring in patients with cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* Patients who visited the hospital emergency room due to cardiac arrest within 60 months after Institutional Review Board (IRB) approval
* Patients with Glasgow Coma Scale (GCS) less than 8 points after spontaneous circulation recovery
* Patients who are 18 years old or older
* Patients who underwent targeted temperature management (TTM)
* Patients who showed good neurological outcomes with CPC 1-2 points after evaluating the prognosis on days 10-14 after ROSC

Exclusion Criteria:

* Under 18 years of age
* cardiac arrest cause is trauma
* Patients who have not undergone targeted temperature management
* Patients treated with extracorporeal membrane oxygenation (ECMO)
* Patients who were not able to undergo SNSB testing
* Patients who could not be followed up until 6 months after ROSC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For subjects who survived after out-of-hospital cardiac arrest, the prognosis was evaluated 10-14 days after ROSC using CPC. For CPC 1-2, neurological prognosis was evaluated as good, and for CPC 3-5, neurological prognosis was evaluated as poor. Only cases of CPC 1-2 between 10 and 14 days after ROSC were included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in cognitive impairment | at 10-14 days, 3 months, and 6 months after return of spontaneous circulation
  Through the Seoul Neuropsychological Screening Battery (SNSB), attention, language and related functions, visuospatial function, memory, frontal lobe and executive function, and other related functions can be assessed. The test is conducted by a specialist clinical psychologist for 1 hour and 30 minutes to 2 hours, and the results are analyzed by Professor Oh Eung-Seok, a neurologist.

CONTACTS AND LOCATIONS:
Overall Officials: Jung Soo Park, MD.Phd, Study Chair — (35015) Chungnam National University Hospital, 282 Munhwa-ro, Jung-gu, Daejeon
Locations (1):
- 박정수, Daejeon, Seo-gu, South Korea

IPD SHARING:
Plan to Share IPD: No
There are no plans to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Result] Cronberg T, Greer DM, Lilja G, Moulaert V, Swindell P, Rossetti AO. Brain injury after cardiac arrest: from prognostication of comatose patients to rehabilitation. Lancet Neurol. 2020 Jul;19(7):611-622. doi: 10.1016/S1474-4422(20)30117-4. PMID 32562686
- [Result] Bronnick K, Evald L, Duez CHV, Grejs AM, Jeppesen AN, Kirkegaard H, Nielsen JF, Soreide E. Biomarker prognostication of cognitive impairment may be feasible even in out-of hospital cardical arrest survivors with good neurological outcome. Resuscitation. 2021 May;162:396-402. doi: 10.1016/j.resuscitation.2021.02.025. Epub 2021 Feb 22. PMID 33631291
- [Result] Moulaert VR, Verbunt JA, van Heugten CM, Wade DT. Cognitive impairments in survivors of out-of-hospital cardiac arrest: a systematic review. Resuscitation. 2009 Mar;80(3):297-305. doi: 10.1016/j.resuscitation.2008.10.034. Epub 2008 Dec 30. PMID 19117659
- [Result] Elliott VJ, Rodgers DL, Brett SJ. Systematic review of quality of life and other patient-centred outcomes after cardiac arrest survival. Resuscitation. 2011 Mar;82(3):247-56. doi: 10.1016/j.resuscitation.2010.10.030. Epub 2011 Jan 8. PMID 21216080